CLINICAL TRIAL: NCT01912235
Title: Arginine Synthesis in Healthy Adult Humans: Does Proline or Glutamate Provide the 5-Carbon Chain?
Brief Title: Arginine Synthesis in Healthy Adult Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Emeritus Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02/02/2010
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Arginine synthesis; 15N2 arginine, 1-13C Glutamine, 2-15N Glutamine, 15N Proline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Study 1: 2-15N glutamine (Active Comparator): To determine the contributions make by glutamine to the provision of nitrogen for ornithine, citrulline and arginine syntesis in adults.
  Interventions: Other: 2-15N glutamine
- Test Study 2: 15N2 arginine &15N proline (Active Comparator): administration of 15N2 arginine &15N proline to measure arginine and proline flux
  Interventions: Other: 15N2 arginine and 15N proline
- Study Test 3: 1-13C glutamine (Active Comparator): to determine to contribution of glutamine to the carbon skeleton of ornithine, citrulline and arginine in adults.
  Interventions: Other: 1-13C glutamine

INTERVENTIONS:
Other: 2-15N glutamine — Glutamine with N15 isotope tracer
  Arms: Test Study 1: 2-15N glutamine
Other: 15N2 arginine and 15N proline — Arginine and Proline isotope tracers
  Arms: Test Study 2: 15N2 arginine &15N proline
Other: 1-13C glutamine — Glutamine carbon isotope tracer
  Arms: Study Test 3: 1-13C glutamine

SUMMARY:
Arginine synthesis in mammals is a complex process involving at least 8 enzymes and intracellular and interorgan transfer of substrates.

The investigators have shown in our neonatal studies that there is no conversion of glutamate to arginine but proline label appears in ornithine, citrulline and arginine. It is clear therefore that arginine is synthesized in human neonates from proline.

In adults the source of the carbon backbone is less clear.

DETAILED DESCRIPTION:
Through a series of test in healthy adults using tandem mass spectrometry with carbon labeled GLN and nitrogen labeled PRO to determine the dietary source for the carbon chain of ORN, CIT and ARG. Additionally, using Nitrogen labeled GLN, we will identify the source of the nitrogen atoms in these amino acids.

Using guanidino - 15N2 arginine, 1-13C Glutamine, 2-15N Glutamine and 15N Proline we will be able to:

1. determine the flux of arginine and proline in healthy adult volunteers
2. determine and compare the flux of carbon and nitrogen labeled glutamine
3. demonstrate whether glutamine or proline provides the carbon backbone for ornithine, citrulline and arginine in adults.
4. the source of the N atoms in ornithine, citrulline and arginine.

ELIGIBILITY:
Inclusion Criteria:

* 5 men of average weight 80 kg will be studied
* healthy, with no know disease of liver, and/or kidney
* weight stable

Exclusion Criteria:

* weith loss or gain over the last three months
* on medications known to affect amino acid metabolism
* known liver, kidney disease condition

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Blood Isotope Levels | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pencharz, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Tomlinson C, Rafii M, Ball RO, Pencharz PB. Arginine can be synthesized from enteral proline in healthy adult humans. J Nutr. 2011 Aug;141(8):1432-6. doi: 10.3945/jn.110.137224. Epub 2011 Jun 15. PMID 21677074
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/21677074